CLINICAL TRIAL: NCT05645029
Title: Antimicrobial Activity and Clinical Performance of Glass Ionomer Cement Modified With Chlorhexidine and Titanium Dioxide in Primary Molars: A Randomized Clinical Trial
Brief Title: Evaluation of Glass Ionomer Cement Modified With Chlorhexidine and Titanium Dioxide in Primary Molars (RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariem Wassel, assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec IR072203
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Dental Caries in Children
MeSH Terms: interventions — glass ionomer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- glass ionomer-chlorhexidine (Experimental)
  Interventions: Other: glass ionomer-chlorhexidine
- glass ionomer -titanium dioxide powder. (Experimental)
  Interventions: Other: glass ionomer-titanium dioxide powder
- glass ionomer (Active Comparator)
  Interventions: Other: glass ionomer

INTERVENTIONS:
Other: glass ionomer-chlorhexidine — chlorhexidine will be added to glass ionomer
  Arms: glass ionomer-chlorhexidine
Other: glass ionomer-titanium dioxide powder — titanium dioxide will be added to glass ionomer
  Arms: glass ionomer -titanium dioxide powder.
Other: glass ionomer — glass ionomer will be used without any additives
  Arms: glass ionomer

SUMMARY:
to investigate the effect of modifying GIC with different formulations on the antibacterial activity and clinical performance in reference to unmodified glass ionomer restorative materials.

DETAILED DESCRIPTION:
The study will be a randomized clinical trial, with a 1:1:1 allocation ratio and parallel arms that will enroll children from the outpatient clinic of pediatric dentistry department, Ain shams University Blinding: Enrolled children, assessors and statistician will be blinded. Randomization: block randomization with blocks of 6. A maximum of 2 primary molars per patient will receive the same treatment.

Allocation concealment: Allocation will be done just before placement of a restoration to avoid performance bias during the cavity preparation. The envelope will be only checked after cavity preparation when the filling material will be chosen

Groups Teeth will be randomly allocated to 3 groups all groups will receive the same cavity preparation and then a different restoration.

* Group A: glass ionomer powder will be mixed with chlorhexidine
* Group B: glass ionomer will be mixed with titanium dioxide powder.
* Group C: will be the positive control, glass ionomer with no additives

Sample Size The sample size: A total number is 39 (13 in each group) is calculated using Epicalc program version 1.02 assuming a power of 80 % and alpha=0.05. The sample size is based on percentage of success of ART restorations at 9 months follow up (GIC with chlorhexidine and GIC with miswak) was 60% and 90%, respectively.13

Intervention:

Teeth will be randomly allocated to the three groups. Care givers and patients involved will be informed about the study procedures, an informed consent form and assent will be obtained. Group A: Conventional glass ionomer cement (Fuji IX, GC, Tokyo, Japan) will be used and modified by incorporating CHX diacetate (0.5% wt) into the powder of the glass ionomer (Fuji IX, GC, Tokyo, Japan) Group B: Conventional glass ionomer cement (Fuji IX, GC, Tokyo, Japan) will be used and modified by incorporating titanium dioxide (3% wt) in glass-based powder component of the GIC.

Group C: Conventional glass ionomer

Cavity preparation and baseline sampling Rubber dam will be placed for isolation of the designated teeth. A step wise caries removal technique will be employed28. Access to the cavity was created using a high-speed dental handpiece fitted with a Meisinger (Hager & Meisinger - Germany) round diamond bur (801G-16) , and all the caries on the lateral walls, caries in the dentine-enamel junction and undermined enamel was removed.

Using a discoid Lascod (Lascod S.p.A Italy) excavator (#1) elective removal of superficial soft necrotic dentine was attempted, leaving behind demineralized wet, leathery dentine centrally on the pulpal wall (Leathery dentine is characterized by being removed in flakes by the excavator) 8,27 A different sterile excavator of the size will be used with very light pressure to take a sample of dentine from the center of the cavity floor center, the sample will be inserted in a brain heart infusion tube and sent to the microbiology lab within 1 hour then added to the culture to measure the bacterial load for the baseline sample by measuring the colony forming units (CFU) 29,30. Blood agar will be used to quantify the total bacterial count, while mitis-salivaris -bacitracin agar will be used to selectively quantify S.mutans.

After cavity preparation, an endodontic file will be used to record the depth of the cavity to aid with the re-entry, and then the operator will reveal the patient's group by opening an envelope. GC cavity conditioner" (GC Japan) will be applied to the cavity walls for 20 seconds leaving the floor unconditioned then the material will be packed into the cavity using a ball burnisher and pressed into it with a petroleum jelly covered gloves for 30 s (press finger technique). Then the excess material will be removed using a carver, and occlusion will be checked and adjusted, then Equia coat varnish (GC Japan) will be applied.

Follow-up The patients will be recalled at 6 and 9 months for clinical performance evaluation by the USPHS evaluation criteria (table 1). Visual and clinical inspection with 3.5x magnification will be done with the help of a sharp explorer by a blinded secondary investigator.

ELIGIBILITY:
Inclusion Criteria:

* The teeth will be primary molars selected from patients presented to the outpatient clinic that are

  * Healthy patients.
  * Children having at least one primary molar with only occlusal caries having dentine lesions (ADA caries classification system mostly 1 or 2 please check)
  * Dentine caries must be apparent visually or radiographically

Exclusion Criteria:

.Teeth with pulp involvement, those suffering from pain, irreversible pulpits or pulp necrosis.

* Patients with history of active para-functional oral habits, xerostomia.
* Patients who will have difficulties in cooperating

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
clinical performance | 9 months
  the clinical performance of different restorations will be evaluated by USPHS evaluation criteria

SECONDARY OUTCOMES:
antibacterial effect | 9 months
  bacterial count reduction will be assessed in dentin

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry .Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No